CLINICAL TRIAL: NCT04765826
Title: Comparison Between Systemic Steroids, Topical Steroids, or Calcineurin Inhibitors With Mini Punch Grafting in Treatment of Stable Non-segmental Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maha, principle investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mahaderma
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Vitiligo
Keywords: vitiligo; mini punch grafting; oral mini pulse steroids; topical treatment
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose oral steroids (Experimental): (20 patients) will receive high dose oral mini pulse steroids (dexamethasone 5 mg on two consecutive weekly days for 3 months).
  Interventions: Procedure: Autologous mini punch grafting
- low dose oral steroids (Experimental): (20 patients) will receive low dose oral mini pulse steroids (2.5mg dexamethasone on two consecutive weekly days for 3 months
  Interventions: Procedure: Autologous mini punch grafting
- topical treatment (Experimental): (20 patients) chosen lesions of comparable size and location in each patient in this group will receive either; super potent topical steroids once every other day, Tacrolimus ointment twice daily for 3 months, or nothing to serve as a control.
  Interventions: Procedure: Autologous mini punch grafting

INTERVENTIONS:
Procedure: Autologous mini punch grafting — All the medications will be administered for 3 months prior to surgery in addition to twice-weekly NB-UVB sessions following its standard protocol.and all patients will continue the treatment till the end of the follow up period Only stable non-responsive or poorly responsive patients (<25% according to VASI score vitiligo area severity index) and image J measurement during the 1st 3 months phase will be included.
  . Chosen lesions in all included patient's groups will undergo mini-punch grafting Mini punch grafting: Skin grafts will be harvested from the anesthetized (local inﬁltration of 2% lignocaine) donor site (the anterolateral aspect of the thigh, using 1mm sterile disposable punches. The grafts obtained will be placed in the slots made by removing the vitiliginous skin using 1mm punches at the recipient site

SUMMARY:
The study to compare the outcomes of mini punch grafting in patients with resistant stable non-segmental vitiligo already on narrowband ultraviolet B and receiving either no additional medication , systemic mini pulse (high and low dose) steroids, topical superpotent steroids once every other day , or daily tacrolimus ointment .in terms of the extent of repigmentation , frequency of reactivation and side effects.

DETAILED DESCRIPTION:
Vitiligo, a depigmenting skin disorder, is characterized by the selective loss of melanocytes, which in turn leads to pigment dilution or loss in the affected areas of the skin. Vitiligo reportedly affects 0.5% to 2% of the world's population, without a clear preference for race or sex. Vitiligo is clinically classified into two main clinical patterns: nonsegmental and segmental. Dermoscopy facilitates the diagnosis of vitiligo .and can be used to assess the evolution of the stage of the disease (stability, progression, repigmentation) as well as the response to treatment. Stability of vitiligo refers to the arrest of disease activity, in terms of the absence of new lesions, no extension of pre-existing lesions, and an absence of Koebner's phenomenon among other features. The duration of stability is a matter of debate, ranging from as little as six months to as long as two years Recent studies have indicated that skin lesions observed in vitiligo tend to recur in the same places where they were found before treatment. This phenomenon is explained by the presence of a recently described subset of memory T cells known as cluster of differentiation( CD8 + )resident memory T cells (TRM) in lesional vitiligo patient skin and a role in disease maintenance and relapse following treatment has been suggested. Thus, the use of immunosuppressants/modulators could ameliorate their activity hence playing a role in stabilizing or treating the disease. . They could also improve the results of surgical options utilized in stable vitiligo refractory to medical treatments including tissue grafts (full-thickness punch, split-thickness, and suction blister grafts), cellular grafts (autologous melanocyte cultures and non-cultured epidermal cellular grafts. In addition to cultured epidermal suspensions and hair follicle transplantation These immune-modulators include: systemic and topical corticosteroids, a topical calcineurin inhibitor, and phototherapy

ELIGIBILITY:
Inclusion Criteria:

Patients of either gender aged more than 18 years old, with stable resistant non-segmental vitiligo will be included.

Stability is defined in terms of:

1. Absence of new lesions or extension of preexisting lesions prior to presentation for the last 6 months.
2. Absence of koebner phenomenon, confetti lesions or hypopigmented lesions, or lesions with ill-defined borders during this same time period.
3. Absence of activity signs by dermoscopic examination which includes :

   * Ill-defined or trichrome border.
   * Micro-Koebner's phenomenon.
   * Tapioca sago appearance.
   * Starburst appearance.
   * Comet tail appearance.
   * Altered pigment network. Resistance to treatment is defined in terms of not responding or those responding poorly to administered treatment (<25% repigmentation according to VASI score) over the last 3 months, especially in patients having lesions on glabrous skin or those with lesions showing leukotrichia.

Exclusion Criteria:

Cases of active, the progressive disease having any of the features of activity listed above during the last 6 months.

Patients with regressive disease showing evidence of repigmentation under administered therapy.

Patients with segmental vitiligo or vitiligo affecting more than 70% body surface area.

Patients with associated autoimmune diseases or any other comorbidity. Patients with a tendency towards hypertrophic scars or keloid formation. Pregnant and breast-feeding females. Patients with psychological instability and unrealistic expectations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of repigmentation and signs of reactivation | 9 months
  assessment of repigmentation will be performed by two blinded dermatologists using a 5-point scale
  ;grade 0(no repigmentation),grade 1(1%-5%),grade 2(6%-25%),grade3(26%-50%),grade4(51%-75%),grade5(76%-100%)
Evaluation of type, pattern and extent of re pigmentation | 9 months
  serial photography will be done to evaluate type, pattern and extent of re pigmentation

CONTACTS AND LOCATIONS:
Overall Officials: Carmen brahiem farid amin, Ph.D, Study Director — Assistant professor of dermatology faculty of medicine .University of Alexandria; Ai Ahmed fouad El Eriny, Ph.D, Study Director — Professor of dermatology faculty of medicine .University of Alexandria; Eman Hamed El Morsy, Ph.D, Study Director — Professor of dermatology faculty of medicine .University of Alexandria
Locations (1):
- Alexandria faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No